CLINICAL TRIAL: NCT05145374
Title: Multivariable Artificial Pancreas to Detect and Mitigate the Effects of Unannounced Physical Activities and Acute Psychological Stress
Brief Title: Multivariable Artificial Pancreas: Detecting and Mitigating Unannounced Physical Activity and Acute Psychological Stress
Status: Recruiting | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Illinois Institute of Technology (Other)
Responsible Party: Principal Investigator, Laurie Quinn, Clinical Professor, University of Illinois at Chicago
Other Study IDs: 2021-0415
Record Dates: First submitted 2021-11-21; First posted 2021-12-06 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Type 1 Diabetes
Keywords: Physical Activity; Psychological Stress; Artificial Pancreas; Sleep; Stress
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Stress, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stressful Stimuli: Participation in meal, exercise, sleep activities alone or in combination with stressful stimuli.

SUMMARY:
The objective of this proposal is to demonstrate a viable, functionally integrated multivariable artificial pancreas (mvAP) that will address meal, physical activity (PA) and acute psychological stress (APS) challenges without any manual inputs to better regulate glucose levels of people with diabetes. Acute psychological stress and many other forms of PA besides planned exercise can affect blood glucose levels and cause challenges to maintaining euglycemia for people with type 1 diabetes mellitus (T1DM). Various PA and APS affect the metabolism and sensitivity to insulin in different ways. Hence, their types, intensities and durations, and their individual and concurrent presence must be detected in order to determine the optimal insulin administration. The mvAP approach provides a well-integrated and user-friendly technology with minimal burden on the user and mitigates the effects of unexpected PA and APS inducements. Twenty subjects with type 1 diabetes (ages 18-60) who use insulin pumps enrolled in this study. The study will take place at the UIC-College of Nursing Diabetes and Exercise Laboratory. The protocol will include 1 screening visit and 5 sessions at the laboratory. The primary activities at each meeting will include: (1) screening; (2) measurement of peak exercise capacity; (3) estimation of maximal strength from submaximal strength tests; (4) Trier Social Stress Test; (5) submaximal bouts of aerobic and resistance exercise, and activities of daily living with and without stress (e.g., mental calculations, video games). These activities will be included visit 3, 4 and 5 as appropriate. In addition, subjects will perform activities at home include: housekeeping chores, stationary bike (if available); treadmill (if available); walking; and light weights (if available). Periodically, the research assistant will call the subject during these times and ask them to perform stress-inducing activities while performing the activity. The stress inducing activities will include mental challenges such as a mathematical computation while performing the activity. The subjects will be called at home 3-5 times during the study. The fully automated algorithm will be tested in a home setting, however, the methodology will be developed and approved for testing later in the study.

DETAILED DESCRIPTION:
The development of an artificial pancreas (AP) has gained considerable progress over the last decade. The goal of AP systems is to develop a device that will provide insulin on demand in response to blood glucose levels in the same manner as the own pancreas. The first generation of AP systems, the hybrid closed-loop AP, collects data from continuous glucose monitoring (CGM) devices and relies on manual user inputs for mitigating the effects of meals and physical activities. The objective of this proposal is to demonstrate a viable, functionally integrated multivariable artificial pancreas (mvAP) that will address meal, physical activity (PA) and acute psychological stress (APS) challenges without any manual inputs to better regulate glucose levels of people with diabetes. Acute psychological stress and many other forms of PA besides planned exercise can affect blood glucose levels and cause challenges to maintaining euglycemia for people with type 1 diabetes mellitus (T1DM). Various PA and APS affect the metabolism and sensitivity to insulin in different ways. Hence, their types, intensities and durations, and their individual and concurrent presence must be detected in order to determine the optimal insulin administration. The mvAP approach provides a well-integrated and user-friendly technology with minimal burden on the user and mitigates the effects of unexpected PA and APS inducements. The objective of this proposal is to demonstrate a viable, functionally integrated mvAP that will address meal, PA and APS challenges without any manual inputs to better regulate glucose levels of people with T1DM. Our hypothesis is that a new generation multivariable AP that incorporates real-time detection and determination of the characteristics of PA and APS and mitigation of their effects by automatic control will be more effective in improving glucose control in people with T1DM. Additionally, this technology will be safer compared to APs based exclusively on CGM data, by reducing the number and duration of hypoglycemic and hyperglycemic events. Such mvAP systems can only be developed by using a sophisticated multivariable approach that uses real-time information from CGMs and physiological variables obtained from wearable devices worn in free-living daily life. It is proposed to build on this framework a fully automated mvAP technology that will mitigate meal, PA and APS challenges, including unexpected and unplanned events. The specific aims of the proposed research are: Aim 1. To develop the mvAP algorithms and modules that identify various types of physical activities, acute psychological stress episodes, their concurrent presence and their characteristics in real time. Aim 2a: To conduct open-loop studies in clinic and in free living to expand the types and intensities of PA and APS inducements, to enrich our database with data collected during activities of daily living (alone or coupled with APS), including unplanned spontaneous PA and APS events. Aim 2b:To extend our multivariable glucose-insulin-physiological variables simulator (mGIPsim) for in silico studies of the mvAP for simulating APS inducements and their effects on glucose levels and physiological variable outputs of the simulator. Aim 3: To conduct clinical experiments with the second generation mvAP in clinical settings and in free living to assess the performance of our fully-automated mvAP in closed-loop operation. At this time, IRB approval for Aim 1, 2a and 2b has been obtained. Aim 3 will be conducted at a later date. The clinical studies will take place at the University of Illinois at Chicago (UIC)-College of Nursing and at the subjects' home. The protocol will include 1 screening visit and 5 sessions at the laboratory. Subjects will wear a CGM and both Empatica and Actigraph wristbands throughout the study. The primary activities at each meeting will include: (1) screening; (2)estimation of maximal exercise capacity from sub-maximal exercise tests (bicycle and treadmill); (3) estimation of maximal strength from sub-maximal strength tests; (4) sub-maximal bouts of aerobic and resistance exercise; (5) use of Socially Evaluated Cold Pressor Test; (6) driving simulation; (7) resistance exercise, and activities of daily living with and without stress (e.g., mental calculations, video games); (8) use of GoPro/Dash Cam during driving (if appropriate) and questionnaires.These activities will be included in visit 3, 4 and 5 as appropriate. In addition, subjects will perform activities at home including: housekeeping chores, stationary bike (if available); treadmill (if available); walking; and light weights (if available) and a sleep monitor (Z-Machine Insight+). Periodically, the research assistant will call the subject during these times and ask them to perform stress-inducing activities while performing the activity. The stress inducing activities will include mental challenges such as a mathematical computation while performing the activity. The subjects will be called at home 3-5 times during the study. The fully automated algorithm will be tested in a home setting. Once the methodology is refined, Institutional Review Board (IRB) approval for the Aim 3 will be obtained.

ELIGIBILITY:
Inclusion Criteria:

Men and Women with T1DM

Insulin pump users

Exclusion Criteria:

* Metabolic instability as evidenced by hospitalizations for diabetes or other diabetes-related complications (e.g., diabetic ketoacidosis and hypoglycemic seizures) within the preceding three months;
* Severe macrovascular disease, as evidenced by severe peripheral artery disease; history of myocardial infarction, heart failure, thromboembolic disease, or unstable angina; uncontrolled hypertension; abnormal resting EKG;
* Maximal exercise stress test with significant brady/tachy arrhythmia, ectopic beats, bundle branch block, or signs of acute ischemia;
* Severe microvascular disease as evidenced by history of vision-threatening proliferative or non-proliferative retinal disease; kidney disease;
* Any uncontrolled non-musculoskeletal condition that would limit the subject's ability to participate in the exercise program (e.g., chronic obstructive airways disease);
* Musculoskeletal conditions such as neurological or orthopedic conditions affecting lower limb strength and mobility (e.g., stroke; insensitive foot);
* Pregnancy;
* Documented medical condition or physical impairment that is judged by the health care practitioner to contraindicate exercise.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Men and Women with Type 1 Diabetes
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of Glucose Concentration | 2 years
  • Glucose concentration (mg/dl) will be measured by: Continuous Glucose Monitor

CONTACTS AND LOCATIONS:
Overall Officials: Ali Cinar, Principal Investigator — Illinois Institute of Technology
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sevil M, Rashid M, Hajizadeh I, Askari MR, Hobbs N, Brandt R, Park M, Quinn L, Cinar A. Discrimination of simultaneous psychological and physical stressors using wristband biosignals. Comput Methods Programs Biomed. 2021 Feb;199:105898. doi: 10.1016/j.cmpb.2020.105898. Epub 2020 Dec 17. PMID 33360529
- [Background] Sevil M, Rashid M, Maloney Z, Hajizadeh I, Samadi S, Askari MR, Hobbs N, Brandt R, Park M, Quinn L, Cinar A. Determining Physical Activity Characteristics from Wristband Data for Use in Automated Insulin Delivery Systems. IEEE Sens J. 2020 Nov;20(21):12859-12870. doi: 10.1109/jsen.2020.3000772. Epub 2020 Jun 8. PMID 33100923
- [Background] Rashid M, Samadi S, Sevil M, Hajizadeh I, Kolodziej P, Hobbs N, Maloney Z, Brandt R, Feng J, Park M, Quinn L, Cinar A. Simulation Software for Assessment of Nonlinear and Adaptive Multivariable Control Algorithms: Glucose - Insulin Dynamics in Type 1 Diabetes. Comput Chem Eng. 2019 Nov 2;130:106565. doi: 10.1016/j.compchemeng.2019.106565. Epub 2019 Sep 2. PMID 32863472
- [Background] Turksoy K, Hajizadeh I, Hobbs N, Kilkus J, Littlejohn E, Samadi S, Feng J, Sevil M, Lazaro C, Ritthaler J, Hibner B, Devine N, Quinn L, Cinar A. Multivariable Artificial Pancreas for Various Exercise Types and Intensities. Diabetes Technol Ther. 2018 Oct;20(10):662-671. doi: 10.1089/dia.2018.0072. Epub 2018 Sep 6. PMID 30188192
- [Background] Brandt R, Park M, Wroblewski K, Quinn L, Tasali E, Cinar A. Sleep quality and glycaemic variability in a real-life setting in adults with type 1 diabetes. Diabetologia. 2021 Oct;64(10):2159-2169. doi: 10.1007/s00125-021-05500-9. Epub 2021 Jun 17. PMID 34136937